CLINICAL TRIAL: NCT00178386
Title: Comparison of Educational Services and Outcomes for Patients Treated for Childhood Cancer and Brain Tumor in Facilities With and Without Educational Liaison Services.
Brief Title: Comparison of Educational Services and Outcomes for Patients Treated for Childhood Cancer
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, OJ Sahler, Professor, University of Rochester
Other Study IDs: 10309
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Cancer; Brain Tumor
Keywords: cancer; education; learning; brain tumor; school
MeSH Terms: conditions — Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to evaluate some educational outcomes of children treated for childhood cancer.

DETAILED DESCRIPTION:
The aim of this telephone survey was to test the efficacy of systemic educational program services in improving school outcomes as compared to hospitals who provide educational liaison services in an ad hoc manner.Data from this study will be used to help secure funding to surther investigate the broader use of educational liaison services.

ELIGIBILITY:
Inclusion Criteria:

* must have had childhood cancer or brain tumor and been diagnosed between 1994-2001 and at least 6 years of age at diagnosis.
* must have been treated at Golisano Children's Hospital or Children's Hospital of Pittsburgh

Exclusion Criteria:

* less than 6 years of age

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2004-09; Primary Completion 2005-09 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Wissler, MS, Principal Investigator — University of Rochester; Robert B Noll, PhD, Principal Investigator — University of Pittsburgh; Olle Jane Z Sahler, MD, Principal Investigator — University of Rochester; Georgia Beyer, MS, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - University of Rochester Golisano Children's Hospital, Rochester, New York
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania